CLINICAL TRIAL: NCT03087162
Title: Once Daily Dose Dexlansoprazole Levofloxacin Based Quadruple Therapy for Helicobacter Pylori Eradication: A Randomized Controlled Study
Brief Title: Once Daily Dose Dexlansoprazole Quadruple Therapy for Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Parin siriwat, Fellowship of Gastroenterology Unit, Ramathibodi Hospital, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Psiriwat
Record Dates: First submitted 2017-02-09; First posted 2017-03-22 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: H Pylori Eradication
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Once daily dose dexlansoprazole (Experimental): Group 1 Dexlansoprazole 60 mg by oral once daily for 14 days (Levofloxacin 500 mg by oral once daily for 14 days Amoxicillin 1000 mg by oral bid for 14 days Bismuth 1048 mg by oral bid for 14 days)
  Interventions: Drug: Dexlansoprazole 60 mg once daily
- Twice daily dose dexlansoprazole (Active Comparator): Group 2 Dexlansoprazole 60 mg oral bid 14 Days (Levofloxacin 500 mg od oral 14 Days Amoxicillin 1000 mg bid oral 14 Days Bismuth 1048 mg bid oral 14 Days)
  Interventions: Drug: Dexlansoprazole 60 mg once daily

INTERVENTIONS:
Drug: Dexlansoprazole 60 mg once daily — Once daily dose dexlansoprazole(Dexlansoprazole(60) OD) in experimental arm and Twice daily dose dexlansoprazole(Dexlansoprazole(60) 1 BID) in active arm
  Other Names: dexilant

SUMMARY:
New drug regimen for Helicobacter pylori eradication, the investigators compare once daily dose dexlansoprazole levofloxacin based quadruple therapy and twice daily dose dexlansoprazole levofloxacin quadruple therapy for helicobacter pylori eradication.

DETAILED DESCRIPTION:
Once daily dose dexlansoprazole should be non inferior to twice daily dose in the eradication of Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 year-patient
2. Diagnosed as positive Helicobacter Pylori testing by any of the following methods:

   * Rapid urease test or Histology
3. Inform consent

Exclusion Criteria:

1. Previous history of Helicobacter pylori eradication
2. Contraindications or allergic reactions to the study drugs
3. Previous gastric surgery or advanced gastric cancer or other malignancy or other severe concurrent diseases
4. Decompensated Liver cirrhosis or chronic kidney disease (GFR< 30)
5. Mental disorders or alcohol or drug addiction
6. Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Eradication rate (percentage) | Jan17-Nov17, Total 11 months
  Compare eradication rate of helicobacter pylori between 2 groups

SECONDARY OUTCOMES:
To compare drug compliance | jan17-Nov17, Total 11 months
  The investigators measure drug compliance between 2 groups, The investigators consider more than 85% of taking medications is a good compliance.
To compare drug adverse event | jan17-Nov17, Total 11 months
  The investigators measure adverse events as
  1. Nausea/Vomiting
  2. Abdominal pain/Abdominal discomfort/Abdominal Bloating
  3. Diarrhea/ Constipation
  4. Taste distortions
  5. Headache/Dizziness
  6. Rash/Itching/Drug allergy, Any symptoms occur new onset during taking medications, The investigators consider as an adverse events of an experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Akrawit Pulsombat, Doctor, Study Director — Ramathibodi Hospital
Locations (1):
- Parin siriwat, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03087162/Prot_000.pdf